CLINICAL TRIAL: NCT03129711
Title: Patient Satisfaction and One Year Clinical Evaluation of Glazed IPS Empress CAD Versus Glazed Celtra Duo Ceramic Laminate Veneers
Brief Title: Patient Satisfaction of Glazed IPS Empress CAD Versus Glazed Celtra Duo Ceramic Laminate Veneers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omnia Mohammed Wafik, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1691985
Record Dates: First submitted 2017-04-24; First posted 2017-04-26 (Actual); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Tooth Discoloration; Tooth Fractures
MeSH Terms: conditions — Tooth Discoloration; Tooth Fractures

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- glazed Celtra Duo (Experimental): zirconia reinforced lithium silicate glass ceramic is infiltrated with 10% zirconia by weight, producing zirconia reinforced lithium silicate ceramic
  Interventions: Other: glazed Celtra Duo
- Glazed IPS Empress CAD (Active Comparator): glazed Leucite based glass ceramics ,Its a glass ceramic which is etchable and proved to have good esthetics if used for laminate veneers
  Interventions: Other: IPS Empress CAD

INTERVENTIONS:
Other: glazed Celtra Duo — zirconia reinforced lithium silicate
  Arms: glazed Celtra Duo
Other: IPS Empress CAD — Standard etchable glass ceramic for laminate veneers
  Other Names: Leucite based
  Arms: Glazed IPS Empress CAD

SUMMARY:
The most frequent reason for failure of laminate veneers made of glass ceramics (feldspathic, leucite based and lithium silicate based ceramics) was fracture of the ceramic, Therefore, ceramic materials that have higher fracture resistance, especially for patients suffering from abnormal occlusion, are needed.

DETAILED DESCRIPTION:
IPS Empress CAD is a leucite glass-ceramic of the SiO2-Al2-O3-K2O material systems with leucite crystal ranging from 5 to 10 µm in size. The leucite crystals increase the material strength and interferes with crack propagation, while the fracture energy is absorbed by the crystalline phase. The resistance and flexural strength (160 Mpa) is improved by the difference in the coefficient of thermal expansion between the glass phase and the crystalline phase and the cooling process following sintering phase.

CELTRA DUO: is a new generation of glass ceramic material. With the aid of a new manufacturing process, the glass ceramic is infiltrated with 10% zirconia by weight, producing zirconia reinforced lithium silicate ceramic (ZLS). The material is characterized by a unique homogenous structure with fine grains that provides excellent material quality and consistency, high strength properties and long term performance. In addition, the material offers satisfying processing characteristics which can be milled and polished easily. After milling the restorations are shaded correctly shaded, with no need for crystallization step 10. The milled restorations have a flexural strength of 210 MPa. After stain and glaze firing the restoration will exhibit a flexural strength up to 370 MPa.

ELIGIBILITY:
Inclusion Criteria:

* All subjects are required to be

  1. From 18-50 years old, be able to read and sign the informed consent document.
  2. Physically and psychologically able to tolerate conventional restorative procedures
  3. have no active periodontal or pulpal diseases, have teeth with good restorations
  4. Patients with teeth problems indicated for laminate veneer:

     1. Discoloration
     2. Fracture not involving more than 50% enamel loss
     3. Mild malposition
     4. Diastema
     5. Enamel fluorosis
     6. Stained or defective restorations
  5. Willing to return for follow-up examinations and evaluation

Exclusion Criteria:

* 1. Patients in the growth stage with partially erupted teeth 2. Patient with fractured teeth of more than 50% enamel loss 3. Patients with poor oral hygiene and motivation 4. Pregnant women's 5. Patient with post and core endodontically treated teeth 6. Psychiatric problems or unrealistic expectations 7. Lack of opposite occluding dentition in the area intended for restoration 8. Patients involved in contact sports 9. Teeth with deep discoloration

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2018-08 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
fracture resistance | 1 year
  scores

IPD SHARING:
Plan to Share IPD: Undecided